CLINICAL TRIAL: NCT05678036
Title: Effects on Mortality and Clinical Course of a Patient's Choice Model for Opioid Maintenance Treatment for Opioid Dependence - Evaluation of a System Enabling a Large Expansion of Treatment Providers and Treatment Access
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Anders C Håkansson, Professor, Region Skane
Other Study IDs: Evaluation of OMT choice model
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Opioid Dependence; Overdose
Keywords: opioid dependence; opioid maintenance treatment; methadone; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose | interventions — Opiate Substitution Treatment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Opioid maintenance treatment — A reform dramatically expanding access to opioid maintenance treatment (with methadone or buprenorphine) in the region.

SUMMARY:
Opioid dependence, for example involving addiction to injected or inhaled heroin or similar compounds, is associated with high mortality, typically from opioid overdose, and causes major physical and mental health complications, social problems and crime. Opioid maintenance treatment (OMT) has proven effective in opioid dependence. In 2014, a patient's choice reform in Skåne county, Sweden, was introduced and led to a vast extension of OMT in the region, including a large number of treatment providers and high access to treatment. Still, opioid-related mortality in the region remains high. While patients' access to treatment has been increased, the content and nature of treatment in the present system has been questioned. The present system, which dramatically altered treatment conditions and access for OMT in this region, has never been formally evaluated in any large-scale study. This study aims to assess clinical course of patients receiving OMT before and during the patient choice reform system, and effects on the extent and nature of opioid-related mortality in the region.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in opioid maintenance treatment in Skåne region.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in opioid maintenance treatment in Skåne region since 2014
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | study inclusion through 2022
  Mortality and cause of death
Hospitalization for substance use disorder treatment | study inclusion through 2022
  Hospitalization for substance use disorder treatment

SECONDARY OUTCOMES:
Mental health disorder | study inclusion through 2022
  Occurrence of a mental health disorder diagnosis aparts from opioid dependence in diagnosis and prescription drug registers
Physical disorder | study inclusion through 2022
  Occurrence of a physical disorder diagnosis aparts from opioid dependence in diagnosis and prescription drug registers

CONTACTS AND LOCATIONS:
Overall Officials: Anders Håkansson, PhD, Principal Investigator — Region Skåne
Locations (1):
- Malmö Addiction Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No